CLINICAL TRIAL: NCT03247140
Title: An Open Label, Randomized, Single-dose, 4-period Cross-over Study to Compare the Pharmacokinetics and Safety Following Administration of JLP-1401 and Coadministration of Rosuvastatin and Telmisartan/Amlodipine in Healthy Adult Volunteers
Brief Title: The PK Characteristics of the Co-administration of Rosuvastatin and Telmisartan/Amlodipine and JLP-1401 in Healthy Male Volunteers Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1401-101-PK
Record Dates: First submitted 2017-07-28; First posted 2017-08-11 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Hypertension With Dyslipidemia
MeSH Terms: interventions — Telmisartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (JLP-1401) (Experimental): JLP-1401(Telmisartan 80 mg, amlodipine 10 mg, rosuvastatin 20 mg)
  Interventions: Drug: JLP-1401; Drug: Telmisartan/Amlodipine, Rosuvastatin
- Group II(Telmisartan/Amlodipine, Rosuvastatin) (Experimental): Twinsta(Telmisartan 40 mg, amlodipine 5 mg) 2 tab and Crestor(rosuvastatin 20 mg)
  Interventions: Drug: JLP-1401; Drug: Telmisartan/Amlodipine, Rosuvastatin

INTERVENTIONS:
Drug: JLP-1401 — Administration of JLP-1401(Telmisartan/Amlodipine/Rosuvastatin)
Drug: Telmisartan/Amlodipine, Rosuvastatin — Administration of Temlisartan/Amlosipine(Twinsta®) and Rosuvastatin(Crestor®)

SUMMARY:
The PK Characteristics of the Co-administration of Rosuvastatin and Telmisartan/Amlodipine and JLP-1401 in Healthy Male Volunteers Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age is over 19 years Body weight is over 55kg, The result of Body Mass Index(BMI) is not less than 17.5 kg/m2 , no more than 30.5 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
* Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
* Subjects who are allergic to investigational drug.
* Subjects who have a medical history which can affect the clinical trial.
* Systolic BP > 140mmHG or Diastolic BP > 90mmHg)
* AST or ALT > X 2 UNL
* History of drug abuse or positive drug screening.
* Participation in other drug studies within 3 months prior to the drug administration.
* Whole blood donation within 60 days, blood component donation within 30 days or who got transfusion within 30days.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
AUC | 72hr after baseline
  Area under the curve of telmisartan, amlodipine, rosuvastatin at 72 hours after baseline
Cmax | 72 after baseline
  Peak concentration of telmisartan, amlodipine, rosuvastatin at 72 hours after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul Kim, MD., Ph.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No